CLINICAL TRIAL: NCT04996095
Title: The Registry Study of Genetic Alterations of Esophageal Cancer in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TCOG T4221
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; precision medicine
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Tumor Sample(s): One H&E staining slide, and 10-15 tissue slides (4-5 um thickness) for cancer panel.
  2. Details of Tests/Collaborative Test Unit:
     Testing will take place in a certified precision medicine laboratory.
  3. Non-tumor Sample (Blood): Eighteen (18) ml of blood will be collected from the participant: 10 ml in EDTA tube (purple top) and 8 ml in Cell-Free DNA blood collection tube.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol Objectives Establish a platform for sharing integrated database of genetic background, clinical information, and therapeutic outcomes in locally advanced and recurrent/metastatic ESCC.

To enroll a total of 400 ESCC patients with different ages and stages according to the eligibility criteria defined in section 5 and section 6.To perform NGS analysis of ESCC tumor tissues, and correlated with the clinical characteristics and treatment outcomes of ESCC patients.To compare the difference of the genetic and molecular profiles among different age groups of ESCC patients.To reveal the evolution changes of genetic and molecular profiles of ESCC by comparing the difference of genetic and molecular alterations between primary and recurrent ESCC and between locally advanced and metastatic ESCC. 。 Study Method, Procedures, and Implementation Status Sample size: 400 patients with ESCC who fit inclusion criteria and exclusion criteria listed in session 6 of the study proposal.

1. To meet the study object of investigating "the difference of the genetic and molecular profiles among different age groups", a minimum of 75 young ESCC patients (with age of ESCC diagnosis at 20-45 years old) and a minimum of 75 elderly ESCC patients (with age of ESCC diagnosis at ≥ 75 years old) will be recruited.
2. To meet the study object of investigating "the evolution changes of genetic and molecular profiles of ESCC", an approximate of 100 recurrent or metastatic ESCC tumors will be included. Centralized Planning Unit and Assisting Unit: Taiwan Cooperative Oncology Group (TCOG), National Health Research Institutes

DETAILED DESCRIPTION:
Esophageal squamous cell carcinoma (ESCC) is a major histological subtype of esophageal cancer in Asia including Taiwan, with distinct epidemiological, clinical, and pathological features from esophageal adenocarcinoma which is commonly seen in Western countries. For decades, esophageal cancer has ranked as one of top leading causes of cancer-related death in Taiwan. Most ESCC patients are men, and present with locally advanced or metastatic disease at diagnosis. Chemoradiotherapy and surgery are commonly employed in patients with locally advanced ESCC; however, more than half of them would eventually develop disease recurrence or distant metastasis. Chemotherapy is the mainstay of treatment for patients with recurrent and metastatic ESCC; unfortunately, the efficacy of chemotherapy has been limited and unsatisfactory. Even anti-program cell death protein 1 (PD-1)- based immunotherapy has recently become an important treatment modality for advanced ESCC, the prognosis of these patients remains poor with a median survival time around a year. Therefore, a better understanding of this deadly disease is crucial for finding better therapeutic strategies for these patients.

A trend of increasing incidence in young age (less than 45-years-old) has been observed in Taiwan recently. This disease not only could devastate these young patients but also would cause huge financial impact to their families. In one of our previous study focusing on the prognosis of metastatic or recurrent ESCC patients treated with systemic chemotherapy, the investigators found that elderly ESCC patients might have better prognosis than young patients. Additionally, the preliminary data of our recent works suggest that the genetic alterations of ESCC in patients of different age groups might be distinct. However, whether the genetic alterations are significantly different among ESCC patients of different age groups and whether the differences exhibit any prognostic or predictive impact have not yet been systematically investigated.

The investigators thus proposed this multi-center research project to address the fore-mentioned questions by collecting tumor tissues from ESCC patients for next-generation sequencing analysis with a panel of cancer-related genes, and creating a platform for data storage and sharing. The specific aims of this project are (1) to establish the tumor genetic and molecular profiles of ESCC in Taiwan, (2) to compare the difference of the genetic and molecular profiles among different age groups of ESCC patients, and (3) to reveal the evolution changes of genetic and molecular profiles of ESCC. The long-term goals of this study are to help implement personalized therapy, to develop novel therapy, and to improve outcomes of patients with ESCC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Cohort 1 (young ESCC): aged 20 ~ 45 years old; Cohort 2 (reference-age ESCC): aged 46 ~ 74 years old); and Cohort 3 (elderly ESCC): aged 75 years or older.

  2. Pathological reported as squamous cell carcinoma of the esophagus 3. Staged as clinical or pathological stage II to IVA in loco-regional ESCC group (per AJCC Cancer Staging System 8th edition); stage IVB in the metastatic group; or recurrent status (defined as disease recurrence occurring more than 6 months after curative chemoradiotherapy or surgery) in the recurrent group.

  4. Willingness to provide archival or newly obtained tumor tissues for current study proposal.

  5. Life expectancy more than 3 months. 6. Patients fully understand the protocol with the willingness to have regular follow-up.

6.2. Exclusion Criteria

1. Inability to cooperate by providing a complete medical history.
2. No available tumor tissues for genetic testing.
3. Undesirable compliance.
4. Having a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.

Exclusion Criteria:

* 1. Inability to cooperate by providing a complete medical history. 2. No available tumor tissues for genetic testing. 3. Undesirable compliance. 4. Having a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1 ESCC:2.Pathological reported as squamous cell carcinoma of the esophagus 3.Staged as clinical or pathological stage II to IVA in loco-regional ESCC group (per AJCC Cancer Staging System 8th edition); stage IVB in the metastatic group; or recurrent status (defined as disease recurrence occurring more than 6 months after curative chemoradiotherapy or surgery) in the recurrent group.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of Predictive Markers | 5 year
  440 cancer-related genes, 31 fusion genes, 500X coverage and the panel size larger than 1MB

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, MD,PHD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Shang-Hung Chen, Tainan
  - Taiwan Cooperative Oncology Group, National Health Research Institutes, Taipei